CLINICAL TRIAL: NCT03715218
Title: Indian Postpartum Care: A-randomised Trial to Improve Maternal Health Six Weeks After Birth
Brief Title: Impact of Mothers Touch Program to Improve Maternal Health After Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NMP Medical Research Institute (Other)
Collaborators: Warwick Research Services (Other); Mothers Touch Foundation, India (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NMP 0146
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Post Partum Depression; Quality of Life
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mother Touch Program (Experimental): Post natal care provided by trained carer after the birth. 6 weeks of care included massage, special diet, physical and mental relaxations.
  Interventions: Other: Mothers Touch Program
- Usual care Program (Other): Usual care and supervision was provided as usual.
  Interventions: Other: Usual Care Program

INTERVENTIONS:
Other: Mothers Touch Program — Mothers Touch Program with bed rest, Relaxation program to reduce stress, massage for mother and infant, gently physical exercise and special dietary program each week.
  Arms: Mother Touch Program
Other: Usual Care Program — Usual care group had advice, support and educational program delivered by midwife, or physicians.
  Arms: Usual care Program

SUMMARY:
After the child birth most women experience major health issues such as depression, severe fatigue, back pain, perineal pain, mastitis, urinary or faecal incontinence, sexual problems and relationship problems with partners. That all lead to poorer emotional and mental health and factors contributing isolation, exhaustion and physical health problems.

'Sava Mahina (6-week period) is a traditional practice for postpartum women in India, which include special diet, lifestyle and supportive care. The current multicenter randomized controlled trial (RCT) aims to evaluate outcomes of Indian postpartum care on women.

ELIGIBILITY:
Inclusion Criteria:

* Primigravida
* Healthy pregnancy
* Consent to participate

Exclusion Criteria:

* Mental Health diagnosis
* Severe depression or psychosis
* Substance abuse

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2018-01-21 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-08-12 (Actual)

PRIMARY OUTCOMES:
Change in Post-natal depression | 6 weeks following child birth
  Changes were assessed using Edinburgh Postnatal Depression scale

SECONDARY OUTCOMES:
Change in Quality of Life | 6 weeks following child birth
  Quality of life was measured using Short Form-36

CONTACTS AND LOCATIONS:
Overall Officials: Rekha Chaudhari, Study Chair — Mothers Touch Foundation, India; Neha Sharma, Principal Investigator — Warwick Research Services; Sangram Birje, Study Director — Mothers Touch Foundation, India; Aparna Chaudhari, Study Director — Mothers Touch Foundation, India
Locations (1):
- NMP Medical Reserach Institute, Jaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yonemoto N, Nagai S, Mori R. Schedules for home visits in the early postpartum period. Cochrane Database Syst Rev. 2021 Jul 21;7(7):CD009326. doi: 10.1002/14651858.CD009326.pub4. PMID 34286512